CLINICAL TRIAL: NCT01742715
Title: Three Methods for Best PEEP Determination Compared With PEEP Determination Guided by Adult Respiratory Distress Syndrome (ARDS) Network, a Crossover Study.
Brief Title: Three Methods for Best PEEP Determination Compared With PEEP Determination Guided by Adult Respiratory Distress Syndrome (ARDS) Network
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0156-12-WOMC
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-10

CONDITIONS: ARDS
Keywords: ARDS; Lung compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEEP by Best oxygenation (Experimental): Set Positive End Expiratory Pressure (PEEP) at 25 cmH2O with fixed driving pressure that will result in delivery of a fixed Tidal Volume (TV) of 6ml/kg Ideal Body Weight (IBW). fraction of inspired oxygen (FiO2) is set to 60%.
  Then decrease PEEP in steps of 4 cmH2O every 10 min until PEEP of 5 cm H2O is reached. In each step static compliance of respiratory system and lung compliance will be measured along with arterial blood gas (ABGs), and hemodynamic parameters such as cardiac output and mixed venous O2 saturation. Best or optimal PEEP will be defined as the PEEP below which PaO2 /FIO2 falls by at least 20%. If at least 20% Partial Oxygen tension (PaO2) PaO2 /FIO2 decrement is not obtained, then PEEP that will result in the highest PaO2 will be selected.
  Interventions: Other: PEEP by Best oxygenation; Other: PEEP by Best Compliance; Other: PEEP by Esophageal pressure
- PEEP by Best Compliance (Experimental): In this group assessment begins with measuring intrinsic PEEP by an expiratory hold. Thereafter, plateau pressures will be recorded after a 0.5-sec inspiratory pause.
  Applied PEEP will be increased by steps of 4 cm H2O, after each incremental step the patient will be observed for 10 minutes to allow for lung unit recruitment and equilibration. Plateau pressure will be measured after each incremental step of PEEP. Applied PEEP will be increased sequentially by 4 cm H2O increments until peak inspiratory pressure of 50 cm H2O, or plateau pressure of 40 cm H2O reached, or hypotension or decrease of 20% in cardiac output is observed.
  Interventions: Other: PEEP by Best oxygenation; Other: PEEP by Best Compliance; Other: PEEP by Esophageal pressure
- PEEP by Esophageal pressure (Experimental): Upon patient recruitment Esophageal balloon will be inserted and esophageal / pleural pressure will be measured. Thereafter, Inspiratory pressures and PEEP will be adjusted according to well established criteria. Inspiratory pressure and PEEP will be adjusted to achieve the best lung compliance possible while not exceeding transpulmonary end Inspiratory pressure of 25 to 30 cm H2O, and at the same time maintaining a positive transpulmonary end expiratory pressure of not more than 5 cm H2O.
  Interventions: Other: PEEP by Best oxygenation; Other: PEEP by Best Compliance; Other: PEEP by Esophageal pressure

INTERVENTIONS:
Other: PEEP by Best oxygenation — Set PEEP at 25 cmH2O with fixed driving pressure that will result in delivery of a fixed Tidal Volume (TV) of 6ml/kg (IBW). FiO2 is set to 60%.
  Then decrease PEEP in steps of 4 cmH2O every 10 min until PEEP of 5 cm H2O is reached. In each step static compliance of respiratory system and lung compliance will be measured along with ABGs, and hemodynamic parameters such as cardiac output and mixed venous O2 saturation. Best or optimal PEEP will be defined as the PEEP below which PaO2 /FIO2 falls by at least 20%. If at least 20% PaO2 /FIO2 decrement is not obtained, then PEEP that will result in the highest PaO2 will be selected.
  Other Names: PEEP determined by Best oxygenation approach.
Other: PEEP by Best Compliance — In this group assessment begins with measuring intrinsic PEEP by an expiratory hold. Thereafter, plateau pressures will be recorded after a 0.5-sec inspiratory pause.
  Applied PEEP will be increased by steps of 4 cm H2O, after each incremental step the patient will be observed for 10 minutes to allow for lung unit recruitment and equilibration. Plateau pressure will be measured after each incremental step of PEEP. Applied PEEP will be increased sequentially by 4 cm H2O increments until peak inspiratory pressure of 50 cm H2O, or plateau pressure of 40 cm H2O reached, or hypotension or decrease of 20% in cardiac output is observed.
Other: PEEP by Esophageal pressure — Upon patient recruitment Esophageal balloon will be inserted and esophageal / pleural pressure will be measured. Thereafter, Inspiratory pressures and PEEP will be adjusted according to well established criteria. Inspiratory pressure and PEEP will be adjusted to achieve the best lung compliance possible while not exceeding transpulmonary end Inspiratory pressure of 25 to 30 cm H2O, and at the same time maintaining a positive transpulmonary end expiratory pressure of not more than 5 cm H2O.

SUMMARY:
To compare the best Positive End Expiratory Pressure (PEEP) as determined by one of three commonly used clinical approaches for best PEEP determination, with PEEP guided by the ARDS network algorithm.

DETAILED DESCRIPTION:
The determination of optimal level of Positive End Expiratory Pressure (PEEP) in patients with acute hypoxemic respiratory pressure remains elusive and controversial.

Several approaches with different algorithms exist. Among them, Low PEEP algorithm approach and High PEEP algorithm approach. These approaches are characterized by a generalized application of certain level of PEEP according to a predefined algorithm. However, these algorithms fail to account for inter-individual variations between patients with different diseases and with different severities of the same underlying process. Therefore, we advocate for an individualized application of PEEP. Whereby, PEEP will be determined individually for each patient based on familiar and well established physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

20 Man and women older than 18 years will be recruited. Patients with acute respiratory failure of any cause who are mechanically ventilated according to the ARDS network recommendations will be considered for inclusion to the study.

To be included in the study a prerequisite of high peak Inspiratory pressure (plateau pressure of 25 to 30 cmH2O) has to be present, and at least one of the following four severity inclusion criteria has to be met.

1 - Low Total Respiratory system compliance (CT), defined as less than 50ml/cmH2O. 2 - PaO2 /FIO2 ratio of less than 300. 3 - Need for a PEEP greater than 10 cmH2O to maintain arterial oxygen saturation (SaO2) of > 90%.

4 - carbon dioxide partial pressure (PCO2) over 60 mmHg, or PH less than 7.2 that is attributed to respiratory acidosis.

Exclusion Criteria:

Patients with any of the following will be excluded from the study. Previous lung or chest wall surgery, previous esophageal surgery, known Achalasia or any other esophageal motility or spasm disorder, presence of chest thoracostomy tube, and any significant chest wall abnormality such as kyphoscoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Oxygenation (defined by partial O2 pressure divided by Fractional inspired Oxygen tension or P/F ratio) | 2 hours
  oxygenation (defined by partial O2 pressure divided by Fractional inspired Oxygen tension or P/F ratio)

SECONDARY OUTCOMES:
Lung compliance (defined by Tidal Volume divided by Inspiratory transpulmonary pressure) | 2 hours
  Lung compliance (defined by Tidal Volume divided by Inspiratory transpulmonary pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, M.D., Principal Investigator — Wolfson MC
Locations (1):
- E. Wolfson MC, Holon, Israel